CLINICAL TRIAL: NCT00618007
Title: A Phase 2, Randomized, Double-Blind, Placebo-Controlled, Parallel Group Study To Evaluate The Efficacy And Safety Of 12-Week Administration Of PF-00734200 To Subjects With Type 2 Diabetes Mellitus And Insufficient Glycemic Control On Metformin Treatment
Brief Title: Effect of PF-00734200 in Subjects With Type 2 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A7941006
Record Dates: First submitted 2008-02-05; First posted 2008-02-18 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — gosogliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 30 mg QD (Experimental)
  Interventions: Drug: PF-00734200 30 mg QD
- 20 mg QD (Experimental)
  Interventions: Drug: PF-00734200 20 mg QD
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-00734200 30 mg QD — 30 mg QD
  Arms: 30 mg QD
Drug: PF-00734200 20 mg QD — 20 mg QD
  Arms: 20 mg QD
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
To determine the effect of PF-00734200 on HbA1c in type 2 diabetic subjects receiving metformin

ELIGIBILITY:
Inclusion Criteria:

Men or women between 18-80 years of age with poorly controlled Type 2 diabetes

Exclusion Criteria:

Type 1 or secondary forms of diabetes Currently using insulin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 289 (Actual)
Dates: Start 2008-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
HbA1c | 12 weeks

SECONDARY OUTCOMES:
Fasting Glucose | 12 weeks
Fasting Insulin | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (71):
- United States (64):
  - Pfizer Investigational Site, Birmingham, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Litchfield Park, Arizona
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Artesia, California
  - Pfizer Investigational Site, Cerritos, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Greenbrea, California
  - Pfizer Investigational Site, Huntington Beach, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, National City, California
  - Pfizer Investigational Site, Roseville, California
  - Pfizer Investigational Site, Valley Village, California
  - Pfizer Investigational Site, West Covina, California
  - Pfizer Investigational Site, DeFuniak Springs, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, New Port Richey, Florida
  - Pfizer Investigational Site, Ocala, Florida
  - Pfizer Investigational Site, Pinecrest, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Idaho Falls, Idaho
  - Pfizer Investigational Site, Indianapolis, Indiana
  - Pfizer Investigational Site, Wichita, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Scarborough, Maine
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Oxon Hill, Maryland
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Bay City, Michigan
  - Pfizer Investigational Site, Canton, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Jackson, Mississippi
  - Pfizer Investigational Site, Picayune, Mississippi
  - Pfizer Investigational Site, City of Saint Peters, Missouri
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, Elizabeth, New Jersey
  - Pfizer Investigational Site, Trenton, New Jersey
  - Pfizer Investigational Site, Albuquerque, New Mexico
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Marion, Ohio
  - Pfizer Investigational Site, Eugene, Oregon
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Aiken, South Carolina
  - Pfizer Investigational Site, Florence, South Carolina
  - Pfizer Investigational Site, Kingsport, Tennessee
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, El Paso, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Hurst, Texas
  - Pfizer Investigational Site, Odessa, Texas
  - Pfizer Investigational Site, Pearland, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Bennington, Vermont
  - Pfizer Investigational Site, Ettrick, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Virginia Beach, Virginia
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Kenosha, Wisconsin
- Canada (5):
  - Pfizer Investigational Site, Coquitlam, British Columbia
  - Pfizer Investigational Site, Toronto, Ontario
  - Pfizer Investigational Site, Laval, Quebec
  - Pfizer Investigational Site, Pointe-Claire, Quebec
  - Pfizer Investigational Site, Québec, Quebec
- Pfizer Investigational Site, San Juan, Puerto Rico
- Pfizer Investigational Site, Seoul, South Korea

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7941006&StudyName=Effect%20of%20PF-00734200%20in%20subjects%20with%20Type%202%20Diabetes